CLINICAL TRIAL: NCT03393260
Title: Epidemiological Characteristics and Prognosis Factors of Cancer Patients Admitted at French Emergency Departments
Acronym: EPICANCER
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: IRU2017
Record Dates: First submitted 2017-12-20; First posted 2018-01-08 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2019-12

CONDITIONS: Cancer Patients; Emergencies
Keywords: cancer; emergency departments (ED)
MeSH Terms: conditions — Emergencies; Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with cancer or hematological malignancy are susceptible to present acute complications linked to their disease or to their specific treatments (dyspnea, sepsis, coma, hemorrhagic syndrome). Emergency physicians are in first line when these complications arise and have to face with some complex situations in which informations about patient malignancy or prognosis may be lacking. Nowadays, there is very few epidemiological data published concerning how cancer patient use Emergency Departments (EDs) and cancer patient care delivery in the EDs.

Thus, an observational multicenter prospective cross-sectional study is conducted to study the prevalence of cancer patients admitted to French EDs, and to describe the different reasons for cancer patients to seek care in EDs with their prevalence and underscore those linked to cancer or treatment complication

ELIGIBILITY:
Inclusion Criteria:

* adult patients (age >=18 years)
* with active malignancy or a history of cancer in remission within the last 5 years
* being attended in one of the 400 French emergency centers participating in the study during the 3-day study period

Exclusion Criteria:

* opposition to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of 18 years or more with active malignancy or in remission for less than 5 years and being attended in one of the 400 French emergency centers participating in the study during 3 consecutive days will be enrolled
Sampling Method: Non-Probability Sample
Enrollment: 1380 (Actual)
Dates: Start 2018-02-06 (Actual); Primary Completion 2018-02-09 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Reasons for cancer patients to seek care in EDs | 1 day

SECONDARY OUTCOMES:
cancer location | 1 day
hospitalisation rate | 1 day
intensive care unit (ICU) admission | 7 days
ICU mortality | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Peyrony, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Saint Louis, Paris, France

REFERENCES:
- [Derived] Peyrony O, Fontaine JP, Trabattoni E, Nakad L, Charreyre S, Picaud A, Bosc J, Viglino D, Jacquin L, Laribi S, Pereira L, Thiriez S, Paquet AL, Tanneau A, Azoulay E, Chevret S, Initiatives de Recherche Aux Urgences Iru-Sfmu Research Group. Cancer Patients' Prehospital Emergency Care: Post Hoc Analysis from the French Prospective Multicenter Study EPICANCER. J Clin Med. 2021 Mar 9;10(5):1145. doi: 10.3390/jcm10051145. PMID 33803366